CLINICAL TRIAL: NCT05206552
Title: The Correlation Between Maternal Infant Bonding , Pain and Postpartum Depression a Prospective Observational Cohort Study
Brief Title: The Correlation Between Maternal Infant Bonding, Pain and Postpartum Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, prinicipal investigator, Rabin Medical Center
Other Study IDs: 0514-21
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Maternal Care Patterns
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients above the age of 18: Study participants will include women after labour whom gave birth to a healthy neonate at 37 weeks with the ability to comply with study requirments
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Maternal - Infant bonding questionnaire. EPDS - Postpartum depression questionnaire

SUMMARY:
The delivery process can be associated with significant maternal pain. which has many long and short term affects.

The aim of our study is to assess whether pain during and after childbirth negatively impacts a mother's attachment to her baby (maternal bonding) and the increases the incidence of postpartum depression.

DETAILED DESCRIPTION:
Delivery is a process that is correlated with maternal pain. The maternal pain can have signifcant long term and short term maternal and neontal impact.

The most common method for pain reilef during delivery is epidural analgesia. Few studies have examined the assocaition between use of epidural analgesia and postpartum depression, with some studies showing a postive correlation and other condricting so.

Maternal bonding is defined as her's emotional state, including maternal feelings towards the infant, it has proven to be the basis for the child's later attachment and sense of self.

A stable and strong bond between mother and child is associated with positive parental behavior and of the child's cognitive and behavioral development, while a unstable maternal infant bond can may lead to long term matenal and infant complications.

The aim of our study is to assess whether pain during and after childbirth negatively impacts a mother's attachment to her baby (maternal bonding) and the increases the incidence of postpartum depression.

In this study women the day after labor will be approched , following obtaining consent will be requested to fill out a the PBO vailadited maternal bonding questtionanire , the valadited EPDS (endinbough postpartum depression questionnaire) and a general questionnaire detailing their demographic , obstetric history and pain levels.

At six weeks postpartum a member of the research team will call the study participant and ask the PBO and EPDS questionnaires to asses the correlation between delivery pain , maternal bonding and postpartum depression,

ELIGIBILITY:
Inclusion Criteria:

*Women whom have given birth at rabin medical center with the ability to follow study requirements.

Exclusion Criteria:

* Women given birth to twins
* Women who's baby was hospitalized
* Women who were treated with magnesium
* Women who's babies were born with congenital malformations

Min Age: 18 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — *Women will be elgible
Study Population: Women whom are the day after labor, who are above the age 18, have given birth to a healthy neonate from 37 weeks of gestation and are able to comply with study requirments
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-01-25 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
Pain verbal numerical score after labor and maternal infant bonding. | 24 hours after labor
  pain levels graded from one to ten will be correlated with maternal infant bonding

SECONDARY OUTCOMES:
Pain verbal numerical score after labor and postpartum depression | 6 weeks after labor
  pain levels graded from one to ten will be correlated with postpartum depression defined as a score of above 10 on the edinbough postpartum depression score questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: sharon orbach-zinger, Principal Investigator — Rabin Medical Center
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shebelsky R, Sadi W, Heesen P, Aber RN, Fein S, Iluz-Freundlich D, Shmueli A, Azem K, Radyan Tamayev I, Binyamin Y, Orbach-Zinger S. The relationship between postpartum pain and mother-infant bonding: A prospective observational study. Anaesth Crit Care Pain Med. 2024 Feb;43(1):101315. doi: 10.1016/j.accpm.2023.101315. Epub 2023 Oct 20. PMID 37865216